CLINICAL TRIAL: NCT04176159
Title: Experimental Research Study About the Effectiveness of a Physiotherapy Program Based on Motor Imagery and Task-oriented Training in Children With Developmental Coordination Disorder
Brief Title: Effectiveness of Motor Imagery and Task-oriented Training in Children With Developmental Coordination Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Moreno Naya (Other)
Responsible Party: Sponsor-Investigator, David Moreno Naya, Principal Investigator, Universidade da Coruña
Organization: Universidade da Coruña (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT29394474
Record Dates: First submitted 2019-11-05; First posted 2019-11-25 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Developmental Coordination Disorder
Keywords: Developmental Coordination Disorder; Task-Oriented Training; Motor Imagery; Physical Therapy
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Intervention Model Description: The subjects will be randomized into 2 groups: an intervention group, which will participate in a program based on the combination of motor imagery and work oriented to the motor task; and a control group, which will carry out their usual school routine.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor imagery and task-oriented training group (Experimental): Two modules. A first module of motor imagery. A second module of task-oriented training and the incorporation of collective activities.
  Interventions: Other: MOTOR IMAGERY AND TASK-ORIENTED TRAINING
- Usual school routines group (No Intervention): Children continue with the usual school routine. Once the study is completed and the corresponding measurements have been made, the subjects included in this group will be subjected to the same program detailed in the intervention, to not deprive them of their benefits.

INTERVENTIONS:
Other: MOTOR IMAGERY AND TASK-ORIENTED TRAINING — The intervention will be divided into two modules. A first module will include activities of activation and relaxation of the body, prediction and sequencing of movement and motor imagery. The second module, task-oriented training, will be divided into analytical work phase (visual coordination, balance, muscular strength, fine motor skills ...), a second phase of integration into specific tasks and, at end, the inclusion of the free (and supervised) practice of a sport.
  The investigators will apply 20 sessions of 40 minutes.
  Arms: Motor imagery and task-oriented training group

SUMMARY:
Experimental study based on the effectiveness of motor imagery and task-oriented training over the motor competence in children with Developmental Coordination Disorder (DCD).

A bilateral hypothesis is assumed for the clinical trial:

* Null hypothesis: physiotherapeutic intervention programs through motor imagery combined with task-oriented training DO NOT modify the parameters of motor competence, anxiety and participation in children susceptible to observation of DCD.
* Alternative hypothesis: physiotherapeutic intervention programs through motor imagery combined with task-oriented training MODIFY the parameters of motor competence, anxiety and participation in children susceptible to observation of DCD.

DETAILED DESCRIPTION:
An experimental and prospective study that will measure changes in motor competence and anxiety levels of school-age children (6 to 12 years old) with suspected presence of Development Coordination Disorder (DCD), before and after participating in a program of physiotherapy based on the combination of motor imagery and task-oriented work developed in their educational center.

A bilateral hypothesis is assumed for the clinical trial:

* Null hypothesis: physiotherapeutic intervention programs through motor imagery combined with task-oriented training DO NOT modify the parameters of motor competence, anxiety and participation in children susceptible to observation of DCD.
* Alternative hypothesis: physiotherapeutic intervention through motor imagery combined with task-oriented training DO modify the parameters of motor competence, anxiety and participation in children susceptible to observation of DCD.

SAMPLE STUDY: the target group will be composed for children of school age, aged between 6 and 12 years (Primary Education), susceptible to diagnosis of Developmental Coordination Disorder.

The recruitment of subjects will be carried out in Primary Education centers framed in the city of A Coruña and its metropolitan area. For this, a first phase of selection or screening will be carried out through the application of a specific questionnaire for the detection of DCD by parents and teachers, and a subsequent analysis of the susceptible subjects through the Movement Assessment Battery for Children, in their second version (MABC-2). The final sample will be composed of those individuals who show a percentile lower than 15 in this battery.

After obtaining informed consent, the subjects will be distributed randomly in 2 groups: an intervention group, with a program based on the combination of motor imagery and motor task oriented training; and a control group, which will carry out their usual school routine. In turn, the groups will be subdivided according to the age group in which the participants are (6-9 years and 10-12 years).

Subsequently, the data of each research subject will be codified.

SAMPLE SIZE:

After the application of the corresponding calculations to the sample size, collecting a 95% confidence interval, a statistical power of 80%, and a loss percentage of 10% of the cases, a minimum sample size of 36 individuals is obtained per each group.

TYPE OF EXPERIMENT AND SELECTED DESIGN: Analytical, longitudinal and prospective research study. Randomized controlled clinical trial with a comparison between an intervention group and a control group.

DATA COLLECT:

1. Personal data: anonymized and coded according to current regulations (RGPD 2016/679 - Europe)
2. Clinical research data:

A. MOTOR COMPETITION: Movement Assessment Battery for Children-Version 2 (MABC-2).

B. ANXIETY LEVEL: Spence Children Anxiety Scale.

C. SATISFACTION, ADHERENCE AND PARTICIPATION: Likert scale.

The data regarding motor competence and anxiety will be taken at the beginning and at the end of the program, as well as in a follow-up measurement that will be carried out 4 weeks later. The satisfaction and adherence scales will be passed only at the end of the study.

All these data will be entered into a specific computer program for later statistical management.

INTERVENTION:

A total of 20 sessions divided into two differential modules will be held. A first module will include activities of activation and relaxation of the body, prediction and sequencing of movement and motor imagery. The second module, of work oriented to the motor task, will be divided into a first phase of analytical work of the altered movement components (visual coordination, balance, muscular strength, fine motor skills ...), a second phase of integration into specific tasks and, at the end, the inclusion of the free (and supervised) sport practice.

STATISTICAL ANALYSIS STRATEGY:

A descriptive study of all the variables will be carried out. Quantitative variables will be expressed as a mean together with their standard deviation value.

Subsequently, randomness, normality and homogeneity tests of variances will be carried out. Depending on the results, the comparison of means will be carried out by parametric or non-parametric means.

All p values <0.05 will be considered statistically significant. The SPSS 23.0 program will be used to proceed with this analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children of school age, aged between 6 and 12, susceptible to the presence of Developmental Coordination Disorder. The sample of participants in the control group will be composed for children with identical characteristics, who will carry out the development of their usual school activity and who will receive the same treatment once the results are obtained.

Exclusion Criteria:

* diagnosed neurological pathology not associated with DCD or any physical or psychological condition that prevents the completion of the proposed intervention.
* absence of authorization of informed consent by a father, mother or legal tutor.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Changes in children´s motor competence | It´s estimated an application time of 20 minutes per evaluation. One application immediately before the intervention and another application immediately after the intervention.
  Changes are measured with the Movement Assessment Battery for Children - Second Version (MABC-2). The final result is composed of scalar scores (from 1 to 19 points), associated with percentiles. Higher scores refer better result.
  The MABC-2 is a standardized test of motor competence assessment aimed at the description and diagnosis of motor problems in children respect to the corresponding development to their age group. The test is presented divided into three age ranges (4-6 years; 7-10 years; 11-16 years). In each range are applied a total of 8 items grouped into three dimensions: manual dexterity, aiming and trapping, and balance (static and dynamic).

SECONDARY OUTCOMES:
Changes in anxiety levels | It´s estimated an application time of 30 minutes per evaluation. One application immediately before the intervention and another application immediately after the intervention.
  Changes are measures with Spence Children´s Anxiety Scale. It consists of 44 items divided into 8 domains: generalized anxiety, panic, separation anxiety, obsessive compulsive disorder, social phobia, fear of physical damage, agoraphobia and compensation of biases.
  Scores range from 0 to 132 points. A higher score identifies greater anxiety.
Satisfaction level: Ad Hoc questionnaire used a Likert scale | A single application of 15 minutes at the eighth week.
  Numerical variables that will be extracted through an Ad Hoc questionnaire used a Likert scale. There are no validated satisfaction scales in this area of research, so it has been decided to develop a scale of its own.
  Scores range from 5 to 35 points. A higher score identifies greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: David Moreno, Principal Investigator
Locations (1):
- CEIP Vales Villamarín, Betanzos, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be published. This protocol is part of a doctoral thesis project linked to the University of A Coruña. The results will be available in the University Repository for free. Subsequently, it will be published in scientific journals and will be available in Research Gate and other similar platforms.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the deposit and defense of the Doctoral Thesis, the data will be available in the Repository of the University of A Coruña for free.
Access Criteria: Initially, the data of the study will be available in the Repository of the University of A Coruña for all those researchers who are interested in the subject, in order to contrast ideas and be useful for future research.

REFERENCES:
- [Background] Biotteau M, Danna J, Baudou E, Puyjarinet F, Velay JL, Albaret JM, Chaix Y. Developmental coordination disorder and dysgraphia: signs and symptoms, diagnosis, and rehabilitation. Neuropsychiatr Dis Treat. 2019 Jul 8;15:1873-1885. doi: 10.2147/NDT.S120514. eCollection 2019. PMID 31371960
- [Background] Gheysen F, Van Waelvelde H, Fias W. Impaired visuo-motor sequence learning in Developmental Coordination Disorder. Res Dev Disabil. 2011 Mar-Apr;32(2):749-56. doi: 10.1016/j.ridd.2010.11.005. Epub 2010 Dec 4. PMID 21131177
- [Background] McHale K, Cermak SA. Fine motor activities in elementary school: preliminary findings and provisional implications for children with fine motor problems. Am J Occup Ther. 1992 Oct;46(10):898-903. doi: 10.5014/ajot.46.10.898. PMID 1463061
- [Background] Wilson PH, McKenzie BE. Information processing deficits associated with developmental coordination disorder: a meta-analysis of research findings. J Child Psychol Psychiatry. 1998 Sep;39(6):829-40. PMID 9758192
- [Background] Blank R, Barnett AL, Cairney J, Green D, Kirby A, Polatajko H, Rosenblum S, Smits-Engelsman B, Sugden D, Wilson P, Vincon S. International clinical practice recommendations on the definition, diagnosis, assessment, intervention, and psychosocial aspects of developmental coordination disorder. Dev Med Child Neurol. 2019 Mar;61(3):242-285. doi: 10.1111/dmcn.14132. Epub 2019 Jan 22. PMID 30671947
- [Background] Blank R. European Academy of Childhood Disability (EACD): Recommendations on the definition, diagnosis and intervention of developmental coordination disorder (pocket version). German-Swiss interdisciplinary clinical practice guideline S3-standard according to the Association of the Scientific Medical Societies in Germany. Pocket version. Definition, diagnosis, assessment, and intervention of developmental coordination disorder (DCD). Dev Med Child Neurol. 2012 Nov;54(11):e1-7. doi: 10.1111/j.1469-8749.2011.04175.x. Epub 2012 Feb 9. No abstract available. PMID 22320659
- [Background] Pratt ML, Hill EL. Anxiety profiles in children with and without developmental coordination disorder. Res Dev Disabil. 2011 Jul-Aug;32(4):1253-9. doi: 10.1016/j.ridd.2011.02.006. Epub 2011 Mar 5. PMID 21377831
- [Background] Smits-Engelsman BC, Blank R, van der Kaay AC, Mosterd-van der Meijs R, Vlugt-van den Brand E, Polatajko HJ, Wilson PH. Efficacy of interventions to improve motor performance in children with developmental coordination disorder: a combined systematic review and meta-analysis. Dev Med Child Neurol. 2013 Mar;55(3):229-37. doi: 10.1111/dmcn.12008. Epub 2012 Oct 29. PMID 23106530
- [Background] Wilson PH, Ruddock S, Smits-Engelsman B, Polatajko H, Blank R. Understanding performance deficits in developmental coordination disorder: a meta-analysis of recent research. Dev Med Child Neurol. 2013 Mar;55(3):217-28. doi: 10.1111/j.1469-8749.2012.04436.x. Epub 2012 Oct 29. PMID 23106668
- [Background] Preston N, Magallon S, Hill LJ, Andrews E, Ahern SM, Mon-Williams M. A systematic review of high quality randomized controlled trials investigating motor skill programmes for children with developmental coordination disorder. Clin Rehabil. 2017 Jul;31(7):857-870. doi: 10.1177/0269215516661014. Epub 2016 Aug 1. PMID 27481937